CLINICAL TRIAL: NCT05267613
Title: A Phase III Study to Assess the Efficacy and Safety of NEXIUM for Maintenance of Healing of Erosive Esophagitis in Pediatric Patients 1 to 11 Years of Age
Brief Title: Endoscopic Evidence of Maintenance of Healing With Oral NEXIUM in Patients 1 to 11 Years Old With Erosive Esophagitis.
Acronym: EE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: IQVIA RDS Inc. (Industry); Calyx (Unknown); Laboratory Corporation of America (Industry); Medidata Solutions (Industry); Thermo Fisher Scientific, Inc (Industry); CISCRP (Industry); Quipment Inc. (Unknown); Little Journey Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9612C09998; 2023-505454-18-00 (Other: EU CT); 2020-002515-21 (EudraCT Number)
Expanded Access: Available
Record Dates: First submitted 2022-01-31; First posted 2022-03-04 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Erosive Esophagitis
Keywords: Erosive Esophagitis; Gastroesophageal Reflux Disease; Healing; Maintenance; Esophagogastroduodenoscopy; Endoscopy; EGD; GERD; GERD in children
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking only applies to the double-blind, randomized maintenance phase of 16 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nexium - high dose (Active Comparator): Arm 1 (High dose = Healing dose)
  Interventions: Drug: Nexium 20mg
- Nexium - Low dose (Active Comparator): Arm 2 (Low dose = ½ healing dose)
  Interventions: Drug: Nexium 10mg

INTERVENTIONS:
Drug: Nexium 20mg — Nexium® (Esomeprazole) gastro-resistant granules for oral suspension 10 or 20 mg taken once daily for 8 weeks, and then 10 or 5 mg taken once daily for 16 weeks.
  Arms: Nexium - high dose
Drug: Nexium 10mg — Nexium® (Esomeprazole) gastro-resistant granules for oral suspension 10 or 20 mg taken once daily for 8 weeks, and then 10 or 5 mg taken once daily for 16 weeks.
  Arms: Nexium - Low dose

SUMMARY:
The aim of the study is to compare the safety and efficacy of two doses of Nexium in maintaining healing of erosive esophagitis in patients 1 to 11 years of age.

DETAILED DESCRIPTION:
Esomeprazole (NEXIUM™) is indicated for the maintenance of healing of endoscopy-verified erosive esophagitis (EE) in children 1 to 11 years of age in a number of countries worldwide, but not in the United States (US). The current study has been designed, in discussions with the Food and Drug Administration (FDA), to further evaluate the safety and efficacy of NEXIUM given as maintenance of healing of EE in children 1 to 11 years of age

Safety assessments will include the monitoring of adverse events throughout the study, clinical laboratory testing (including hematology, clinical chemistry, urinalysis), vital signs (including blood pressure and pulse), and physical examination including weight.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be 1 to 11 years of age
2. Patients must have a clinical history of GERD for at least 3 months before the start of study
3. For the healing phase: Patients must have confirmed presence of EE at endoscopy performed within one week of the start of the healing phase.
4. For the maintenance phase: Patients must have completed the healing phase and have endoscopy-verified healed EE at the 8-week endoscopy visit.
5. Patients must weigh ≥ 10 kg.
6. Patients may be male or female.
7. All postmenarcheal female patients must have a negative pregnancy test (urine) before starting treatment.
8. Sexually active patients must be abstinent or maintain effective contraception from informed consent day up to the last day of study intervention.
9. Patient's guardian must be capable of giving signed informed consent

Exclusion Criteria:

1. Presence of other diseases, such as severe heart, lung, liver, renal, blood, or neurological disease or similar
2. Significant clinical illness within 4 weeks prior to the start of treatment
3. Any conditions that are predicted to require a surgery during the study period (from the day of informed consent to the day of the last scheduled visit)
4. Previous total gastrectomy
5. Anticipated need for concomitant therapy with PPIs (except for the IMPs), H2-receptor antagonists and other drugs outlined in EC#5 after enrollment in this study
6. Participation in another clinical study with an IMP administered in the last 4 weeks before enrollment.
7. Patients with a known hypersensitivity to NEXIUM, or any other PPI, or any of the excipients of the product
8. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
9. Judgment by the Investigator that the patient should not participate in the study if the patient or guardian is unlikely to comply with study procedures, restrictions, and requirements
10. Previous screening, or enrollment and randomization in the present study

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-08-14 (Estimated); Study Completion 2027-09-06 (Estimated)

PRIMARY OUTCOMES:
Presence / absence of Erosive Esophagitis | Week 24 (end of 16-week maintenance phase)
  Presence/absence of Erosive Esophagitis for all patients by assessment of Esophagogastroduodenoscopy at the end of the 16-week maintenance phase

SECONDARY OUTCOMES:
Presence/absence of Erosive Esophagitis | Week 8 (end of healing phase)
  Presence/absence of Erosive Esophagitis for all patients by assessment of Esophagogastroduodenoscopy at the end of the 8-week healing phase
Percentage of days without rescue medication | Week 8 (end of healing phase) and Week 16 (end of maintenance phase)
  The percentage of days without rescue medication during the 8-week healing phase and during the 16-week maintenance phase

CONTACTS AND LOCATIONS:
Locations (45):
- United States (16):
  - Research Site, Mobile, Alabama
  - Research Site, Fontana, California
  - Research Site, Orange, California
  - Research Site, Sacramento, California
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Downers Grove, Illinois
  - Research Site, Carmel, Indiana
  - Research Site, Springfield, Massachusetts
  - Research Site, The Bronx, New York
  - Research Site, Akron, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Knoxville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Milwaukee, Wisconsin
- Argentina (3):
  - Research Site, Córdoba
  - Research Site, Paraná
  - Research Site, Rosario
- Australia (2):
  - Research Site, Clayton
  - Research Site, North Adelaide
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Namur
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Italy (3):
  - Research Site, Messina
  - Research Site, Napoli
  - Research Site, Roma
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Vilnius
- Portugal (5):
  - Research Site, Braga
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Viana do Castelo
- Russia (4):
  - Research Site, Novosibirsk
  - Research Site, Pyatigorsk
  - Research Site, Saint Petersburg
  - Research Site, Tomsk
- Spain (3):
  - Research Site, Badalona
  - Research Site, Santiago de Compostela
  - Research Site, Seville
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Hochiminh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home